CLINICAL TRIAL: NCT04130334
Title: Effects of Corneal Anatomical Match Between Donor and Recipient During DALK Surgery on Final Visual and Refractive Outcomes in Patients With KCN: a Clinical Trial
Brief Title: Effects of Corneal Anatomical Match Between Donor and Recipient During DALK Surgery on Final Visual and Refractive Outcomes in Patients With KCN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10000
Record Dates: First submitted 2019-10-07; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-05

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- horizontal meridian of donor's cornea sutured to horizontal (Active Comparator): horizontal meridian of donor's cornea sutured to horizontal meridian of recipient cornea
  Interventions: Procedure: After mechanical trephination, horizontal meridian of donor's cornea sutured to horizontal meridian of recipient cornea
- horizontal meridian of donor's cornea sutured to vertical (Active Comparator): horizontal meridian of donor's cornea sutured to vertical meridian of recipient cornea
  Interventions: Procedure: : After mechanical trephination, horizontal meridian of donor's cornea sutured to vertical meridian of recipient cornea

INTERVENTIONS:
Procedure: After mechanical trephination, horizontal meridian of donor's cornea sutured to horizontal meridian of recipient cornea — After mechanical trephination, horizontal meridian of donor's cornea sutured to horizontal meridian of recipient cornea
  Arms: horizontal meridian of donor's cornea sutured to horizontal
Procedure: : After mechanical trephination, horizontal meridian of donor's cornea sutured to vertical meridian of recipient cornea — : After mechanical trephination, horizontal meridian of donor's cornea sutured to vertical meridian of recipient cornea
  Arms: horizontal meridian of donor's cornea sutured to vertical

SUMMARY:
Patients with KCN who undergo cornea transplantation divided to 2 groups:

Group1: After mechanical trephination, horizontal meridian of donor's cornea sutured to horizontal meridian of recipient cornea Group 2: After mechanical trephination, horizontal meridian of donor's cornea sutured to vertical meridian of recipient cornea After suture removal, best corrected visual acuity, refractive error, corneal keratometry, irregularity of corneal surface and high order aberration of two groups will compare

ELIGIBILITY:
Inclusion Criteria:

* Patients with KCN who undergo DALK surgery

Exclusion Criteria:

* Penetrating Keratoplasty surgery
* Other corneal diseases
* dystrophies
* Corneal graft rejection

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 14 months
  Snellen chart
graft astigmatism | 14 months
  Topography

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran